CLINICAL TRIAL: NCT02793232
Title: A 3-part Phase 1, Randomized, Double-blind, Sponsor-open, Placebo Controlled Trial To Evaluate The Safety, Tolerability, Food Effect, Pharmacokinetics And Pharmacodynamics Of Pf-06751979 After Oral Administration: Part A - Single Ascending Doses In Healthy Adults; Part B - Multiple Ascending Doses In Healthy Adults; And Part C - Multiple Doses To Older Subjects
Brief Title: Clinical Trial In Healthy Volunteers And Health Elderly Volunteers To Evaluate The Safety, Tolerability And Blood Concentration After Single And Multiple Escalating Oral Doses Of PF-06751979.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B8271004; 2016-000325-39 (EudraCT Number)
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2017-12

CONDITIONS: Healthy Subjects
Keywords: Safety; Tolerability; Pharmacokinetics; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — PF-06751979

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Ascending Dose Crossover (Experimental): Single Ascending Dose in 4-way cross-over design (PF-06751979/Placebo).
  Interventions: Drug: PF-06751979 single dose; Drug: Placebo single dose
- Multiple Ascending Dose (Experimental): Multiple dose administration to Healthy Subjects in parallel cohorts (PF-06751979).
  Interventions: Drug: PF-06751979 multiple ascending dose; Drug: Placebo multiple ascending dose
- Multiple Dose Elderly (Experimental): Multiple dose administration to Healthy Elderly Subjects (PF-06751979). This cohort is optional.
  Interventions: Drug: PF-06751979 multiple dose; Drug: Placebo multiple elderly dose

INTERVENTIONS:
Drug: PF-06751979 single dose — PF-06751979 administered as a single dose suspension in cross-over fashion. Each subject may receive up to 4 study treatments (placebo and up to 3 doses of PF 06751979). The planned dose levels are 200 mg, 400 mg, 700 mg, 200 mg fed (these doses are subject to change based on emerging data).
  Arms: Single Ascending Dose Crossover
Drug: Placebo single dose — Matched Placebo suspension administered as single dose
  Arms: Single Ascending Dose Crossover
Drug: PF-06751979 multiple ascending dose — PF-06751979 suspension administered daily for 14 consecutive days to parallel cohorts. The planned dose levels are mg, 100 mg, 200 mg, 340 mg (these are subject to change based on emerging data).
  Arms: Multiple Ascending Dose
Drug: Placebo multiple ascending dose — Matched placebo suspension administered daily for 14 consecutive days.
  Arms: Multiple Ascending Dose
Drug: PF-06751979 multiple dose — PF-06751979 suspension administered daily for 14 consecutive days. The planned dose level is 340 mg (this is subject to change based on emerging data).
  Arms: Multiple Dose Elderly
Drug: Placebo multiple elderly dose — Multiple dose administration to Healthy Elderly Subjects (Placebo)
  Arms: Multiple Dose Elderly

SUMMARY:
This study will test the safety, tolerability and blood concentrations of single and multiple oral doses of PF-06751979 in health subjects and healthy elderly subjects. PF-06751979 is being developed for the treatment of Alzheimer's disease.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) of PF-06751979 following oral doses in healthy adult and healthy elderly subjects at higher doses than previously administered. Such characteristics will enable the design of future clinical trials in patient population, in the effort to optimize the efficacy of PF-06751979, as well as to establish safety margins in humans. Inclusion of healthy elderly subjects will be optional, but can provide additional safety and tolerability information in the age range of the target population while confirming the PK of PF-06751979 in these subjects for future clinical trials in the Alzheimer's disease patient population.

The Primary Objective is to evaluate the safety and tolerability of single and multiple ascending oral doses of PF-06751979 in healthy adult subjects. Secondary Objectives are to characterize the pharmacokinetics of PF-06751979 in: plasma following single and multiple ascending oral dose administration in healthy adult subjects and urine following multiple ascending oral dose administration in healthy adult subjects. An additional secondary objective is to evaluate the effect of multiple oral doses of PF 06751979 on CSF A-beta fragments in healthy adult subjects.

This study is divided into three parts: Part A - Single ascending doses (SAD) healthy adult subjects (18-55 years); Part B - Multiple ascending doses (MAD) in healthy adult subjects (18-55 years); Part C - Multiple doses (MD) in healthy elderly subjects (60-85 years). Study Parts may be run in a staggered fashion; Part C of the study may commence after satisfactory review of relevant data from Parts A and B.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non childbearing potential and male subjects.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2 (32 kg/m2 for healthy elderly); and a total body weight >50 kg (110 lbs) at Screening.
* Evidence of a personally signed and dated informed consent document indicating that the subject or a legally acceptable representative has been informed of all pertinent aspects of the study.
* Additional criterion for subjects of Japanese descent who may be enrolled in Part B (multiple ascending dose cohorts in healthy subjects): Japanese subjects who have four Japanese grandparents born in Japan.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Unwilling or unable to comply with the Lifestyle Guidelines described in the protocol.
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
* Any severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B8271004&StudyName=A+3-part+Phase+1%2C+Randomized%2C+Double-blind%2C+Sponsor-open%2C+Placebo+Controlled+Trial+To+Evaluate+The+Safety%2C+Tolerability%2C+Food+Effect%2C+Pharmacokinetics+And+Pharmacodynamics+Of+Pf-06751979+After+Oral+Administration%3A++Part+A+-+Single+Ascending+Doses+In+Healthy+Adults%3B+Part+B+-+Multiple+Ascending+Doses+In+Healthy+Adults%3B+And+Part+C+-+Multiple+Doses+To+Elderly+Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B8271004&StudyName=A+3-part+Phase+1%2C+Randomized%2C+Double-blind%2C+Sponsor-open%2C+Placebo+Controlled+Trial+To+Evaluate+The+Safety%2C+Tolerability%2C+Food+Effect%2C+Pharmacokinetics+And+Pharmacodynamics+Of+Pf-06751979+After+Oral+Administration%3A+Part+A+-+Single+Ascending+Doses+In+Healthy+Adults%3B+Part+B+-+Multiple+Ascending+Doses+In+Healthy+Adults%3B+And+Part+C+-+Multiple+Doses+To+Older+Subjects

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was conducted in 3 parts: Part A (4-period cross-over design), Part B and C (single period, parallel design).
Groups:
- Part A- Placebo, PF-06751979: 400 mg, 540 mg, 200 mg Fed: Participants received oral dose of placebo matched to PF-06751979 on Day 1 of intervention period 1 followed by oral dose of PF-06751979 400 milligram (mg) suspension on Day 1 of intervention period 2 followed by oral dose of PF-06751979 540 mg suspension on Day 1 of intervention period 3 followed by an oral dose of PF-06751979 200 mg suspension under fed condition on Day 1 of intervention period 4. A washout period of at least 10 days was maintained between each intervention period. All doses were administered in fasted state except PF-06751979 200 mg Fed. After completion of period 4, participants were followed for 10 days.
- Part A-PF-06751979 200mg,Placebo,PF-06751979 540 mg,200 mg Fed: Participants received oral dose of PF-06751979 200 mg suspension on Day 1 of intervention period 1 followed by oral dose of placebo matched to PF-06751979 on Day 1 of intervention period 2 followed by oral dose of PF-06751979 540 mg suspension on Day 1 of intervention period 3 followed by an oral dose of PF-06751979 200 mg suspension under fed condition on Day 1 of intervention period 4. A washout period of at least 10 days was maintained between each intervention period. All doses were administered in fasted state except PF-06751979 200 mg Fed. After completion of period 4, participants were followed for 10 days.
- Part A-PF-06751979: 200mg, 400mg,Placebo,PF-06751979 200mg Fed: Participants received oral dose of PF-06751979 200 mg suspension on Day 1 of intervention period 1 followed by oral dose of PF-06751979 400 mg suspension on Day 1 of intervention period 2 followed by oral dose of placebo matched to PF-06751979 on Day 1 of intervention period 3 followed by an oral dose of PF-06751979 200 mg suspension under fed condition on Day 1 of intervention period 4. A washout period of at least 10 days was maintained between each intervention period. All doses were administered in fasted state except PF-06751979 200 mg Fed. After completion of period 4, participants were followed for 10 days.
- Part A- PF-06751979: 200 mg, 400 mg, 540 mg, Placebo: Participants received oral dose of PF-06751979 200 mg suspension on Day 1 of intervention period 1 followed by oral dose of PF-06751979 400 mg suspension on Day 1 of intervention period 2 followed by oral dose of PF-06751979 540 mg suspension on Day 1 of intervention period 3 followed by oral dose of placebo matched to PF-06751979 on Day 1 of intervention period 4. A washout period of at least 10 days was maintained between each intervention period. All doses were administered in fasted state. After completion of period 4, participants were followed for 10 days.
- Part B: Placebo; Part C: Placebo: Participants received oral dose of placebo matched to PF-06751979 suspension once daily from Day 1 up to Day 14 in intervention period of 19 days. Participants were followed up to 15 days (up to Day 29) after last dose of study medication.
- Part B: PF-06751979 125 mg; Part C: PF-06751979 125 mg: Participants received oral dose of PF-06751979 125 mg suspension once daily from Day 1 up to Day 14 in intervention period of 19 days. Participants were followed up to 15 days (up to Day 29) after last dose of study medication.
- Part B: PF-06751979 275 mg: Participants received oral dose of PF-06751979 275 mg suspension once daily from Day 1 up to Day 14 in intervention period of 19 days. Participants were followed up to 15 days (up to Day 29) after last dose of study medication.
Period: Period 1-Part A:5 Days; Part B,C:19 Days
Arm/Group | Part A- Placebo, PF-06751979: 400 mg, 540 mg, 200 mg Fed | Part A-PF-06751979 200mg,Placebo,PF-06751979 540 mg,200 mg Fed | Part A-PF-06751979: 200mg, 400mg,Placebo,PF-06751979 200mg Fed | Part A- PF-06751979: 200 mg, 400 mg, 540 mg, Placebo | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Started | 2 | 2 | 2 | 2 | 7 | 12 | 9 | 2 | 8
Completed | 2 | 2 | 2 | 2 | 6 | 12 | 8 | 2 | 8
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Period: Washout Period 1(Part A:at Least 10days)
Arm/Group | Part A- Placebo, PF-06751979: 400 mg, 540 mg, 200 mg Fed | Part A-PF-06751979 200mg,Placebo,PF-06751979 540 mg,200 mg Fed | Part A-PF-06751979: 200mg, 400mg,Placebo,PF-06751979 200mg Fed | Part A- PF-06751979: 200 mg, 400 mg, 540 mg, Placebo | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (Part A: 5 Days)
Arm/Group | Part A- Placebo, PF-06751979: 400 mg, 540 mg, 200 mg Fed | Part A-PF-06751979 200mg,Placebo,PF-06751979 540 mg,200 mg Fed | Part A-PF-06751979: 200mg, 400mg,Placebo,PF-06751979 200mg Fed | Part A- PF-06751979: 200 mg, 400 mg, 540 mg, Placebo | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2(Part A:at Least 10days)
Arm/Group | Part A- Placebo, PF-06751979: 400 mg, 540 mg, 200 mg Fed | Part A-PF-06751979 200mg,Placebo,PF-06751979 540 mg,200 mg Fed | Part A-PF-06751979: 200mg, 400mg,Placebo,PF-06751979 200mg Fed | Part A- PF-06751979: 200 mg, 400 mg, 540 mg, Placebo | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (Part A: 5 Days)
Arm/Group | Part A- Placebo, PF-06751979: 400 mg, 540 mg, 200 mg Fed | Part A-PF-06751979 200mg,Placebo,PF-06751979 540 mg,200 mg Fed | Part A-PF-06751979: 200mg, 400mg,Placebo,PF-06751979 200mg Fed | Part A- PF-06751979: 200 mg, 400 mg, 540 mg, Placebo | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3(Part A:at Least 10days)
Arm/Group | Part A- Placebo, PF-06751979: 400 mg, 540 mg, 200 mg Fed | Part A-PF-06751979 200mg,Placebo,PF-06751979 540 mg,200 mg Fed | Part A-PF-06751979: 200mg, 400mg,Placebo,PF-06751979 200mg Fed | Part A- PF-06751979: 200 mg, 400 mg, 540 mg, Placebo | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 (Part A: 5 Days)
Arm/Group | Part A- Placebo, PF-06751979: 400 mg, 540 mg, 200 mg Fed | Part A-PF-06751979 200mg,Placebo,PF-06751979 540 mg,200 mg Fed | Part A-PF-06751979: 200mg, 400mg,Placebo,PF-06751979 200mg Fed | Part A- PF-06751979: 200 mg, 400 mg, 540 mg, Placebo | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A- Placebo, PF-06751979: 400 mg, 540 mg, 200 mg Fed | Part A-PF-06751979 200mg,Placebo,PF-06751979 540 mg,200 mg Fed | Part A-PF-06751979: 200mg, 400mg,Placebo,PF-06751979 200mg Fed | Part A- PF-06751979: 200 mg, 400 mg, 540 mg, Placebo | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 12 | 9 | 2 | 8 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 2 | 7 | 12 | 9 | 0 | 2 | 38
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
  Male | 2 | 2 | 2 | 2 | 7 | 12 | 9 | 1 | 5 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment emergent were events between first dose of study drug and up to the follow up visit (up to 36 days in Part A, 49 days in Part B and C), that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Part A: Baseline up to 36 days; Part B and C: Baseline up to 49 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Part A: Placebo: All participants who received oral dose of placebo matched to PF-06751979 in either 1 of the 4 intervention periods in Part A of the study. A washout period of at least 10 days was maintained between each intervention period.
- Part A: PF-06751979 200 mg: All participants who received oral dose of PF-06751979 200 mg suspension in either 1 of the 4 intervention periods in Part A of the study. A washout period of at least 10 days was maintained between each intervention period.
- Part A: PF-06751979 400 mg: All participants who received oral dose of PF-06751979 400 mg suspension in either 1 of the 4 intervention periods in Part A of the study. A washout period of at least 10 days was maintained between each intervention period.
- Part A: PF-06751979 540 mg: All participants who received oral dose of PF-06751979 540 mg suspension in either 1 of the 4 intervention periods in Part A of the study. A washout period of at least 10 days was maintained between each intervention period.
- Part A: PF-06751979 200 mg Fed: All participants who received oral dose of PF-06751979 200 mg suspension under fed condition in either 1 of the 4 intervention periods in Part A of the study. A washout period of at least 10 days was maintained between each intervention period.
Arm/Group | Part A: Placebo | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 7 | 12 | 9 | 2 | 8
participants
  AEs | 1 | 3 | 2 | 6 | 4 | 6 | 10 | 8 | 2 | 6
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Abnormal Physical Examinations Findings
Description: Full physical examination included head, ears, eyes, nose, mouth, skin, heart, lung, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. Abnormality in physical examinations was based on investigator's discretion.
Time Frame: Part A: Baseline up to 36 days; Part B and C: Baseline up to 49 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 7 | 12 | 9 | 2 | 8
participants | 1 | 5 | 0 | 0 | 0 | 6 | 8 | 5 | 0 | 4

3. Primary Outcome: Number of Participants With Abnormal Neurological Examinations Findings
Description: The neurological examination included the assessment of higher cortical function, the cranial nerves, motor function, deep tendon reflexes, sensory exam, and coordination and gait. Abnormality in neurological examinations was based on investigator's discretion.
Time Frame: Part A: Baseline up to 36 days; Part B and C: Baseline up to 49 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 7 | 12 | 9 | 2 | 8
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part B and C: Number of Participants With Positive Response on the Columbia Suicide Severity Rating Scale (C-SSRS) at Baseline
Description: C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced following: completed suicide; suicide attempt (response of "Yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("Yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent). In this outcome measure, number of participants with positive response (response of "yes") to suicidal behavior, ideation or any non-suicidal self-injurious behavior, at baseline were reported.
Time Frame: Baseline
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Data for this outcome measure was not planned to be analyzed for Part A, as pre-specified in protocol.
Measure: Number; unit: participants
Arm/Group | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 7 | 12 | 9 | 2 | 8
participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part B and C: Number of Participants With Positive Response on the Columbia Suicide Severity Rating Scale (C-SSRS) at Day 7
Description: C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced following: completed suicide; suicide attempt (response of "Yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("Yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent). In this outcome measure, number of participants with positive response (response of "yes") to suicidal behavior, ideation or any non-suicidal self-injurious behavior, at Day 7 were reported.
Time Frame: Day 7
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 7 | 12 | 9 | 2 | 8
participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part B and C: Number of Participants With Positive Response on the Columbia Suicide Severity Rating Scale (C-SSRS) at Day 14
Description: C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced following: completed suicide; suicide attempt (response of "Yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("Yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent). In this outcome measure, number of participants with positive response (response of "yes") to suicidal behavior, ideation or any non-suicidal self-injurious behavior, at Day 14 were reported.
Time Frame: Day 14
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 7 | 12 | 9 | 2 | 8
participants | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part B and C: Number of Participants With Positive Response on the Columbia Suicide Severity Rating Scale (C-SSRS) at Day 19
Description: C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced following: completed suicide; suicide attempt (response of "Yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("Yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent). In this outcome measure, number of participants with positive response (response of "yes") to suicidal behavior, ideation or any non-suicidal self-injurious behavior, at Day 19 were reported.
Time Frame: Day 19
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 7 | 12 | 9 | 2 | 8
participants | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Criteria for abnormal values of ECG parameters: maximum pulse rate (PR) interval greater than or equal to (>=)300 milliseconds (msec); maximum PR interval increase from baseline (IFB): >=25 percent (%) when baseline was greater than (>)200 msec; or >=50 % when baseline was greater than (>)200 msec, maximum QRS interval >=140 msec and QRS interval IFB: >=50%. QT interval using Fridericia's correction (QTcF) ranges from 450 msec to maximum less than (<)480 msec, less than or equal to (<=) 480 msec to maximum <500 msec and maximum >=500 msec, maximum QTcF interval IFB range from <=30 to <60 msec and maximum >=60 msec. Only categories which included at least 1 participant with abnormality are reported in this outcome measure.
Time Frame: Part A: Baseline up to 36 days; Part B and C: Baseline up to 49 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 7 | 12 | 9 | 2 | 8
participants
  Maximum QTCF Interval: 450 to <480 msec | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Maximum QTCF Interval IFB: <=30 to <60 msec | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

9. Primary Outcome: Part A: Number of Participants With Cardiac Rhythms of Potential Clinical Concern Assessed By Telemetry
Description: In all Periods of Part A, continuous cardiac monitoring was maintained for 8 hours (or longer if considered clinically necessary by the investigator) following dose administration on Day 1. All abnormal cardiac rhythms were recorded and reviewed by the study physician for the presence of rhythms of potential clinical concern.
Time Frame: Day 1
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Data for this outcome measure was not planned to be analyzed for Part B and C, as pre specified in protocol.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Criteria for vital signs abnormalities: systolic blood pressure (SBP) <90 millimeter of mercury (mmHg), diastolic blood pressure (DBP) <50 mmHg, supine pulse rate <40 beats per minute (bpm). Maximum IFB in Supine SBP >=30 mmHg, Maximum decrease from baseline (DFB) in Supine SBP >=30 mmHg, maximum DFB in Supine DBP >=20 mmHg.
Time Frame: Part A: Baseline up to 36 days; Part B and C: Baseline up to 49 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 7 | 12 | 9 | 2 | 8
participants
  Supine SBP: <90 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Supine DBP: <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Supine PR: <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Maximum IFB in Supine SBP: >=30 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Maximum DFB in Supine SBP: >=30 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Maximum DFB in Supine DBP: >=20 mmHg | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1

11. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Abnormalities criteria:hematology(hemoglobin; hematocrit; RBC<0.8*lower limit of normal [LLN]; platelets<0.5*LLN,>1.75*upper limit of normal [ULN]; WBC<0.6*LLN,>1.5*ULN; lymphocytes; neutrophils; basophils; eosinophils; monocytes<0.8*LLN,>1.2*ULN; coagulation(prothrombin ratio>1.1*ULN), liver(bilirubin>1.5*ULN; aspartate aminotransferase; alanine aminotransferase; alkaline phosphatase; gamma GT>0.3*ULN; protein; albumin<0.8*LLN,>1.2*ULN); renal(blood urea nitrogen, creatinine>1.3*ULN; uric acid>1.2*ULN); electrolytes(sodium<0.95*LLN,>1.05*ULN; potassium; chloride; calcium; bicarbonate<0.9*LLN,>1.1*ULN), chemistry(glucose<0.6*LLN,>1.5* ULN); urinalysis(pH <4.5,>8; glucose, ketones, protein, blood, urobilinogen, nitrite, bilirubin, leukocyte, esterase>1; WBC; bacteria>=20, epithelial cells>=6; granular casts, hyaline casts, red cell casts, white cell casts>1; lipids(cholesterol[C], LDL-C>1.3*ULN; HDL-C<0.8*LLN, triglycerides>1.3*ULN); hormones(T4, T3, T4, TSH<0.8*LLN,>1.2*ULN).
Time Frame: Part A: Baseline up to 36 days; Part B and C: Baseline up to 49 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 7 | 12 | 9 | 2 | 8
participants | 6 | 5 | 2 | 3 | 5 | 5 | 11 | 8 | 1 | 7

12. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of PF-06751979
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: Pharmacokinetic (PK) parameter analysis set included all enrolled participants who had at least 1 dose of PF-06751979 and at least of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter | 643.2 (19) | 1436 (10) | 1829 (19) | 630.2 (9)

13. Secondary Outcome: Part A: Area Under the Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of PF-06751979
Description: Area under the plasma concentration-time profile from time zero to the time of last measured concentration (AUClast).
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: PK parameter analysis set included all enrolled participants who had at least 1 dose of PF-06751979 and at least of the PK parameters of interest measured. Data for this outcome measure was not planned to be analyzed for Part B and C, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour per milliliter | 20500 (19) | 41710 (18) | 58190 (14) | 20170 (13)

14. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06751979
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour per milliliter | 22850 (17) | 44980 (17) | 63420 (9) | 23260 (15)

15. Secondary Outcome: Part A: Dose Normalized Maximum Observed Plasma Concentration (Cmax[dn]) of PF-06751979
Description: Cmax(dn) was obtained calculated by dividing Cmax by the exact dose of PF-06751979 (in milligram) administered to a participant.
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: PK parameter analysis set included all enrolled participants who had at least 1 dose of PF-06751979 and at least of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanogram per milliliter) per milligram
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
(nanogram per milliliter) per milligram | 3.218 (19) | 3.592 (10) | 3.387 (19) | 3.154 (9)

16. Secondary Outcome: Part A: Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast[dn]) of PF-06751979
Description: AUClast(dn) was calculated by dividing AUClast by the exact dose of PF-06751979 (in mg) administered to a participant. AUClast was area under the plasma concentration-time profile from time zero to the time of last measured concentration.
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanogram*hour/milliliter) per milligram
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
(nanogram*hour/milliliter) per milligram | 102.6 (19) | 104.2 (18) | 107.9 (14) | 100.9 (13)

17. Secondary Outcome: Part A: Dose Normalized Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUCinf [dn]) of PF-06751979
Description: AUCinf (dn) was calculated by dividing AUCinf by the exact dose of PF-06751979 (in mg) administered to a participant. AUCinf was area under the plasma concentration-time profile from time zero extrapolated to infinite time (0-inf).
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanogram*hour/milliliter) per milligram
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
(nanogram*hour/milliliter) per milligram | 114.1 (17) | 112.4 (17) | 117.6 (9) | 116.4 (15)

18. Secondary Outcome: Part A: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06751979
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 4.00 (17) [2.00 to 6.07] | 3.02 (17) [2.00 to 4.00] | 3.01 (9) [2.00 to 6.02] | 6.00 (15) [4.00 to 8.00]

19. Secondary Outcome: Part A: Plasma Decay Half-Life (t1/2) of PF-06751979
Description: Plasma decay half-life is the time duration for the plasma concentration of PF-06751979 to decrease by one-half of its original concentration.
Time Frame: pre-dose, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 35.20 (8.9731) [2.00 to 6.07] | 34.70 (8.9749) [2.00 to 4.00] | 35.85 (8.1028) [2.00 to 6.02] | 33.38 (6.2474) [4.00 to 8.00]

20. Secondary Outcome: Part A: Apparent Clearance (CL/F) of PF-06751979
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
milliliter per minute | 145.8 (17) [2.00 to 6.07] | 148.3 (17) [2.00 to 4.00] | 142.0 (9) [2.00 to 6.02] | 143.3 (15) [4.00 to 8.00]

21. Secondary Outcome: Part A: Apparent Volume of Distribution (Vz/F) of PF-06751979
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liter | 433.7 (18) [2.00 to 6.07] | 433.0 (19) [2.00 to 4.00] | 431.1 (19) [2.00 to 6.02] | 408.1 (16) [4.00 to 8.00]

22. Secondary Outcome: Part B: Maximum Observed Plasma Concentration (Cmax) of PF-06751979
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose on Day 1; pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose on Day 7; pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: PK parameter analysis set included all enrolled participants who had at least 1 dose of PF-06751979 and at least of the PK parameters of interest measured. Here, number analyzed signifies those participants who were evaluable at specified time points for each arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
nanogram per milliliter
  Day 1 | 442.7 (20) | 983.2 (18)
  Day 7 | 818.7 (19) | 2000 (14)
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 837.6 (16) | 1869 (14)

23. Secondary Outcome: Part B: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06751979
Description: Area under the plasma concentration versus time-curve from time zero to end of dosing interval (AUCtau), where dosing interval was 24 hours.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose on Day 1; pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose on Day 7; pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose on Day 14
Population: Analysis was performed on PK parameter analysis set. Number analyzed= participants evaluable at specified time points for each arm. Data for this outcome measure was not planned to be analyzed for Part A, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
nanogram*hour per milliliter
  Day 1 | 6380 (15) | 13260 (18)
  Day 7 | 13810 (16) | 31210 (14)
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 13990 (14) | 29470 (12)

24. Secondary Outcome: Part B: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06751979
Time Frame: as for outcome 22
Population: PK parameter analysis set included all enrolled participants who had at least 1 dose of PF-06751979 and at least of the PK parameters of interest measured. Here, number analyzed signifies those participants who were evaluable at specified time point for each arm.
Measure: Median (Full Range); unit: hours
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
hours
  Day 1 | 4.00 [2.00 to 6.03] | 4.00 [2.00 to 4.00]
  Day 7 | 3.00 [2.00 to 6.00] | 2.00 [2.00 to 4.00]
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 4.00 [2.00 to 12.00] | 4.00 [2.00 to 4.00]

25. Secondary Outcome: Part B: Dose Normalized Maximum Observed Plasma Concentration (Cmax[dn]) of PF-06751979
Description: Cmax(dn) was obtained calculated by dividing Cmax by the exact dose of PF-06751979 (in mg) administered to a participant.
Time Frame: as for outcome 22
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanogram per milliliter) per milligram
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
(nanogram per milliliter) per milligram
  Day 1 | 3.541 (20) | 3.576 (18)
  Day 7 | 6.549 (19) | 7.272 (14)
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 6.702 (16) | 6.794 (14)

26. Secondary Outcome: Part B: Dose Normalized Area Under the Curve From Time Zero to End of Dosing Interval Tau (AUCtau[dn]) of PF-06751979
Description: Area under the concentration curve from time zero to end of dosing interval (AUCtau), where dosing interval was 24 hours. AUCtau (dn) was calculated by dividing AUCtau by the exact dose of PF-06751979 (in mg) administered to a participant.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanogram*hour/milliliter)/milligram
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
(nanogram*hour/milliliter)/milligram
  Day 1 | 51.04 (15) | 48.21 (18)
  Day 7 | 110.4 (16) | 113.5 (15)
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 111.8 (14) | 107.1 (12)

27. Secondary Outcome: Part B: Apparent Clearance (CL/F) of PF-06751979
Description: as for outcome 20
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose on Day 7; pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
milliliter per minute
  Day 7 | 151.0 (16) | 146.9 (14)
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 149.0 (14) | 155.3 (13)

28. Secondary Outcome: Part B: Minimum Observed Plasma Concentration (Cmin) of PF-06751979
Time Frame: as for outcome 27
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
nanogram per milliliter
  Day 7 | 388.4 (17) | 857.3 (15)
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 390.3 (18) | 868.5 (15)

29. Secondary Outcome: Part B: Peak-to-Trough Ratio of PF-06751979
Description: Peak-to-trough ratio was calculated by dividing Cmax with Cmin of PF-06751979. Cmax was maximum plasma concentration during the dosing interval and Cmin was minimum observed plasma concentration during the dosing interval.
Time Frame: as for outcome 27
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
ratio
  Day 7 | 2.111 (10) | 2.332 (8)
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 2.145 (11) | 2.151 (9)

30. Secondary Outcome: Part B: Observed Accumulation Ratio (Rac) for AUCtau of PF-06751979
Description: Rac for AUCtau for Day 7 was calculated as: AUCtau on Day 7 divided by AUCtau on Day 1. Rac for AUCtau for Day 14 was calculated as: AUCtau on Day 14 divided by AUCtau on Day 1.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
ratio
  Day 7 | 2.165 (9) | 2.355 (15)
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 2.190 (11) | 2.265 (11)

31. Secondary Outcome: Part B: Observed Accumulation Ratio for Maximum Observed Plasma Concentration (Rac Cmax) of PF-06751979
Description: Rac for Cmax on Day 7 was calculated as: Cmax on Day 7 divided by Cmax on Day 1 and Rac for Cmax on Day 14 was calculated as: Cmax on Day 14 divided by Cmax on Day 1, where Cmax was the maximum observed plasma concentration.
Time Frame: as for outcome 22
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 9
ratio
  Day 7 | 1.849 (16) | 2.033 (7)
  Day 14: number analyzed (Participants) | 12 | 8
  Day 14 | 1.892 (14) | 1.923 (9)

32. Secondary Outcome: Part B: Plasma Decay Half-Life (t1/2) of PF-06751979
Description: as for outcome 19
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: PK parameter analysis set included all enrolled participants who had at least 1 dose of PF-06751979 and at least of the PK parameters of interest measured. Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 8
hour | 30.73 (5.7464) [2.00 to 12.00] | 37.79 (7.7261) [2.00 to 4.00]

33. Secondary Outcome: Part B: Apparent Volume of Distribution (Vz/F) of PF-06751979
Description: as for outcome 21
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 12 | 8
Liter | 390.5 (23) [2.00 to 12.00] | 498.3 (27) [2.00 to 4.00]

34. Secondary Outcome: Part C: Maximum Observed Plasma Concentration (Cmax) of PF-06751979
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose on Day 1; pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
nanogram per milliliter
  Day 1 | 377.1 (30) [2.00 to 12.00]
  Day 14 | 879.4 (28)

35. Secondary Outcome: Part C: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06751979
Description: as for outcome 23
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose on Day 1; pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose on Day 14
Population: PK parameter analysis set included all enrolled participants who had at least 1 dose of PF-06751979 and at least of the PK parameters of interest measured. Data for this outcome measure was not planned to be analyzed for Part A, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
nanogram*hour per milliliter
  Day 1 | 5238 (24) [2.00 to 12.00]
  Day 14 | 14750 (23)

36. Secondary Outcome: Part C: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06751979
Time Frame: as for outcome 34
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
hours
  Day 1 | 4.00 (24) [2.00 to 4.03]
  Day 14 | 4.00 [2.00 to 4.03]

37. Secondary Outcome: Part C: Dose Normalized Maximum Observed Plasma Concentration (Cmax[dn]) of PF-06751979
Description: as for outcome 25
Time Frame: as for outcome 34
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanogram per milliliter) per milligram
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
(nanogram per milliliter) per milligram
  Day 1 | 3.019 (30) [2.00 to 4.03]
  Day 14 | 7.035 (28) [2.00 to 4.03]

38. Secondary Outcome: Part C: Dose Normalized Area Under the Curve From Time Zero to End of Dosing Interval Tau (AUCtau[dn]) of PF-06751979
Description: as for outcome 26
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanogram*hour/milliliter)/milligram
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
(nanogram*hour/milliliter)/milligram
  Day 1 | 41.93 (24) [2.00 to 4.03]
  Day 14 | 118.0 (23) [2.00 to 4.03]

39. Secondary Outcome: Part C: Apparent Oral Clearance (CL/F)
Description: as for outcome 20
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
milliliter per minute | 141.4 (23) [2.00 to 4.03]

40. Secondary Outcome: Part C: Minimum Observed Plasma Concentration (Cmin) of PF-06751979
Description: Minimum observed concentration during the dosing interval.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
nanogram per milliliter | 429.9 (23) [2.00 to 4.03]

41. Secondary Outcome: Part C: Peak-to-Trough Ratio of PF-06751979
Description: as for outcome 29
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
ratio | 2.045 (10) [2.00 to 4.03]

42. Secondary Outcome: Part C: Observed Accumulation Ratio (Rac) for AUCtau of PF-06751979
Description: Rac for AUCtau at Day 14 was calculated as: AUCtau on Day 14 divided by AUCtau on Day 1.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
ratio | 2.814 (3) [2.00 to 4.03]

43. Secondary Outcome: Part C: Observed Accumulation Ratio for Maximum Observed Plasma Concentration (Rac Cmax) of PF-06751979
Description: Rac for Cmax on Day 14 was calculated as: Cmax on Day 14 divided by Cmax on Day 1, where Cmax was the maximum observed plasma concentration.
Time Frame: as for outcome 34
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
ratio | 2.332 (7) [2.00 to 4.03]

44. Secondary Outcome: Part C: Plasma Decay Half-Life (t1/2) of PF-06751979
Description: Plasma decay half-life was the time duration for the plasma concentration to decrease by one-half of its original concentration.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
hours | 40.76 (3.9042) [2.00 to 4.03]

45. Secondary Outcome: Part C: Apparent Volume of Distribution (Vz/F) of PF-06751979
Description: as for outcome 21
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part C: PF-06751979 125 mg
Number analyzed (Participants) | 8
Liter | 496.1 (30) [2.00 to 4.03]

46. Secondary Outcome: Part B: Amount of PF-06751979 Excreted Unchanged in Urine Over the Dosing Interval Tau (Aetau)
Description: Aetau was the amount of drug excreted unchanged in urine during the dosing interval tau, where tau was 24 hours.
Time Frame: 0-24 hours on Day 14
Population: PK parameter analysis set =all enrolled participants who had at least 1 dose of PF-06751979 and at least of the PK parameters of interest measured.Here, number of participants analyzed =participants who were evaluable for this outcome measure.Data for this outcome measure was not planned to be analyzed for Part A and C,as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 9 | 8
milligram | 12.93 (38) | 25.93 (28)

47. Secondary Outcome: Part B: Percentage of Dose of PF-06751979 Excreted Unchanged in the Urine Over the Dosing Interval Tau (Aetau%)
Description: Aetau% was calculated as: 100*Aetau/dose. Aetau was the amount of drug excreted unchanged in urine during the dosing interval tau, where tau was 24 hours.
Time Frame: 0-24 hours on Day 14
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose excreated
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 9 | 8
percentage of dose excreated | 10.36 (38) | 9.429 (28)

48. Secondary Outcome: Part B: Renal Clearance of PF-06751979
Description: Renal clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated in urine. It was calculated as amount of drug excreted unchanged in urine during the dosing interval tau (Aetau) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCtau), where dosing interval was 24 hours.
Time Frame: 0-24 hours on Day 14
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute
Arm/Group | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 9 | 8
milliliter per minute | 15.54 (37) | 14.68 (34)

49. Secondary Outcome: Part B: Percent Change From Baseline in Cerebrospinal Spinal Fluid (CSF) Amyloid Beta (ABeta) Fragments
Description: ABeta is the peptide fragment of the amyloid precursor protein. Percent change from baseline in CSF concentration of ABeta fragments (ABeta 1-38, ABeta 1-40, ABeta 1-42, ABeta total, ABeta x-38, ABeta x-40, ABeta x-42, soluble amyloid precursor protein alpha (sAPP-alpha), soluble amyloid precursor protein beta (sAPP-beta) at Day 14 was reported in this outcome measure.
Time Frame: Baseline, Day 14
Population: Pharmacodynamic CSF concentration population: all enrolled and treated participants who had at least 1 measureable CSF ABeta concentration. Number of participants analyzed= participants who were evaluable for this outcome measure. Data for this outcome measure was not planned to be analyzed for Part A and C, as pre specified in protocol.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg
Number analyzed (Participants) | 6 | 12 | 8
percent change
  ABeta 1-38 | -4.223 (0.0669) | -80.324 (0.0472) | -87.935 (0.0579)
  ABeta 1-40 | -10.031 (0.0746) | -85.452 (0.0536) | -92.927 (0.0689)
  ABeta 1-42 | -10.335 (0.0789) | -86.383 (0.0587) | -93.607 (0.0758)
  ABeta x-38 | -12.362 (0.0708) | -82.003 (0.0513) | -90.106 (0.0643)
  ABeta x-40 | -9.785 (0.0673) | -80.998 (0.0478) | -87.622 (0.0591)
  ABeta x-42 | -10.874 (0.0539) | -81.861 (0.0385) | -86.618 (0.0472)
  sAPP-alpha | -8.237 (0.0655) | 58.653 (0.0480) | 81.737 (0.0604)
  sAPP-beta | -5.553 (0.0545) | -81.266 (0.0390) | -84.304 (0.0485)
  ABeta total | -7.911 (0.0492) | -80.116 (0.0348) | -86.523 (0.0428)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: PF-06751979 125 mg; ABeta 1-38: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -79.456, 80% CI 2-sided [-81.56 to -77.11], Standard Error of Mean 0.0819
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: PF-06751979 275 mg; ABeta 1-38: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -87.403, 80% CI 2-sided [-88.80 to -85.84], Standard Error of Mean 0.0887
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: PF-06751979 125 mg; ABeta 1-40: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -83.830, 80% CI 2-sided [-85.65 to -81.78], Standard Error of Mean 0.0905
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: PF-06751979 275 mg; ABeta 1-40: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -92.138, 80% CI 2-sided [-93.15 to -90.98], Standard Error of Mean 0.1041
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: PF-06751979 125 mg; ABeta 1-42: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -84.814, 80% CI 2-sided [-86.64 to -82.74], Standard Error of Mean 0.0971
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: PF-06751979 275 mg; ABeta 1-42: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -92.870, 80% CI 2-sided [-93.85 to -91.74], Standard Error of Mean 0.1114
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B: PF-06751979 125 mg; ABeta x-38: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -79.465, 80% CI 2-sided [-81.69 to -76.96], Standard Error of Mean 0.0870
Statistical Analysis 8: Comparison: Part B: Placebo vs Part B: PF-06751979 275 mg; ABeta x-38: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -88.711, 80% CI 2-sided [-90.06 to -87.18], Standard Error of Mean 0.0963
Statistical Analysis 9: Comparison: Part B: Placebo vs Part B: PF-06751979 125 mg; ABeta x-40: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -78.936, 80% CI 2-sided [-81.11 to -76.52], Standard Error of Mean 0.0824
Statistical Analysis 10: Comparison: Part B: Placebo vs Part B: PF-06751979 275 mg; ABeta x-40: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -86.280, 80% CI 2-sided [-87.82 to -84.55], Standard Error of Mean 0.0899
Statistical Analysis 11: Comparison: Part B: Placebo vs Part B: PF-06751979 125 mg; ABeta x-42: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -79.648, 80% CI 2-sided [-81.36 to -77.78], Standard Error of Mean 0.0664
Statistical Analysis 12: Comparison: Part B: Placebo vs Part B: PF-06751979 275 mg; ABeta x-42: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -84.985, 80% CI 2-sided [-86.34 to -83.50], Standard Error of Mean 0.0715
Statistical Analysis 13: Comparison: Part B: Placebo vs Part B: PF-06751979 125 mg; sAPP-alpha: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = 72.893, 80% CI 2-sided [55.37 to 92.40], Standard Error of Mean 0.0809
Statistical Analysis 14: Comparison: Part B: Placebo vs Part B: PF-06751979 275 mg; sAPP-alpha: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = 98.049, 80% CI 2-sided [75.92 to 122.96], Standard Error of Mean 0.0897
Statistical Analysis 15: Comparison: Part B: Placebo vs Part B: PF-06751979 125 mg; sAPP-beta: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -80.164, 80% CI 2-sided [-81.84 to -78.33], Standard Error of Mean 0.0668
Statistical Analysis 16: Comparison: Part B: Placebo vs Part B: PF-06751979 275 mg; sAPP-beta: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -83.381, 80% CI 2-sided [-84.92 to -81.69], Standard Error of Mean 0.0733
Statistical Analysis 17: Comparison: Part B: Placebo vs Part B: PF-06751979 125 mg; Abeta total: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -78.408, 80% CI 2-sided [-80.06 to -76.62], Standard Error of Mean 0.0602
Statistical Analysis 18: Comparison: Part B: Placebo vs Part B: PF-06751979 275 mg; Abeta total: General linear model with treatment, as the fixed effect and loge(baseline) as covariate; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Percent change from baseline = -85.365, 80% CI 2-sided [-86.57 to -84.05], Standard Error of Mean 0.0653

ADVERSE EVENTS:
Time Frame: Part A: Baseline up to 36 days; Part B and C: Baseline up to 49 days
Arm/Group | Part A: Placebo | Part A: PF-06751979 200 mg | Part A: PF-06751979 400 mg | Part A: PF-06751979 540 mg | Part A: PF-06751979 200 mg Fed | Part B: Placebo | Part B: PF-06751979 125 mg | Part B: PF-06751979 275 mg | Part C: Placebo | Part C: PF-06751979 125 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/12 | 0/9 | 0/2 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/12 | 0/9 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 3/6 | 2/6 | 6/6 | 4/6 | 6/7 | 10/12 | 8/9 | 2/2 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=8) | Part A: PF-06751979 200 mg (N=6) | Part A: PF-06751979 400 mg (N=6) | Part A: PF-06751979 540 mg (N=6) | Part A: PF-06751979 200 mg Fed (N=6) | Part B: Placebo (N=7) | Part B: PF-06751979 125 mg (N=12) | Part B: PF-06751979 275 mg (N=9) | Part C: Placebo (N=2) | Part C: PF-06751979 125 mg (N=8)
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1
Hunger (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 3 | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye movement disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Daydreaming (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.